CLINICAL TRIAL: NCT03876275
Title: Comparative Study of Arthrodeses in One Time by "Single Posterior Approach" and Two-stage Arthrodeses by "Double Anterior and Posterior Approach"
Brief Title: Comparative Study of Arthrodeses by "Single Posterior Approach" and by "Double Anterior and Posterior Approach"
Acronym: ARBORD
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ARBORD
Record Dates: First submitted 2019-03-07; First posted 2019-03-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Spinal Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extended arthrodesis of the spine is indicated in the treatment of deformities. The principle of the intervention is to correct the spinal imbalance and to obtain a fusion of the vertebral segment operated in order to guarantee the durability of this correction, in order to guarantee a functional result the best possible one.

There is a great disparity in the techniques available to obtain this result: as regards the correction of the deformation itself, it is possible to resort to various types of gestures aimed at "freeing" the spine to allow the getting the correction. It may be staged or transpedicular osteotomies or previous releases (staged discectomies). Regarding the arthrodesis itself, this can be obtained by an isolated posterior graft or by a circumferential graft itself performed in a time using interbody cages PLIF type (posterior lumbar interbody fusion) or TLIF (transforaminal interbody fusion) or in two stages by a complementary anterior graft. These are heavy interventions with a high complication rate.

The choice of this or that technique is based on data from the literature and remains at the discretion of the surgeon who makes the surgical indication. However, it has never been possible to compare these different techniques in a prospective study. The few articles comparing the different techniques tend to show that there is no significant difference between the techniques with a higher complication rate for the two-step techniques. However, these are retrospective studies, with all the biases that this implies and despite these results the disparity in surgical indications remains substantial.

The objective of this work is therefore to evaluate, according to an identical protocol, the different surgical techniques for the treatment of spinal deformities associated with a fusion in order to determine the morbidity associated with each of the techniques and if this morbidity is justified by a better functional result at a minimum follow-up of two years.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient operated on an arthrodesis including the sacrum and extending to T11 or greater
* Francophone patient
* Patient not opposing his participation in the research protocol

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing arthrodesis including the sacrum and extending to T11 or greater
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Surgical revision rate | year 2
  Surgical revision rate following double-approach techniques and single posterior approach techniques

SECONDARY OUTCOMES:
duration of the procedure | Day 1
  duration of the procedure
bleeding during the procedure | Day 1
  bleeding volume during the procedure
quality of life questionnary Oswestry v2 | Day 0
  The quality of life questionnary Oswestry v2 before surgery corresponds to the score 0% -20%: Minimal disability; 21%-40%: Moderate Disability; 41%-60%: Severe Disability; 61%-80%: Crippling back pain and 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
quality of life questionnary SF-12 | Day 0
  The quality of life questionnary SF-12 before surgery corresponds to a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
Visual Analog Score for pain | Day 0
  The visual Analog Score for pain before surgery corresponds to a score between 0 to 10.
quality of life questionnary Oswestry v2 | year 1
  The quality of life questionnary Oswestry v2 one year after surgery corresponds to the score 0% -20%: Minimal disability; 21%-40%: Moderate Disability; 41%-60%: Severe Disability; 61%-80%: Crippling back pain and 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
quality of life questionnary SF-12 | year 1
  The quality of life questionnary SF-12 one year after surgery to a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
Visual Analog Score for pain | year 1
  The pain evaluation with Visual analogue scale one year after surgery corresponds to a score between 0 to 10.
quality of life questionnary Oswestry v2 | year 2
  The quality of life questionnary Oswestry v2 two years after surgery corresponds to the score 0% -20%: Minimal disability; 21%-40%: Moderate Disability; 41%-60%: Severe Disability; 61%-80%: Crippling back pain and 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
quality of life questionnary SF-12 | year 2
  The quality of life questionnary SF-12 two years after surgery to a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
Visual Analog Score for pain | year 2
  The pain evaluation with Visual analogue scale two years after surgery corresponds to a score between 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France